CLINICAL TRIAL: NCT00070655
Title: The AMADEUS Trial, A Multicenter, Randomized, Open-label, Assessor Blind, Non-inferiority Study Comparing the Efficacy and Safety of Once-weekly Subcutaneous Idraparinux (SR34006) With Adjusted-dose Oral Vitamin-K Antagonists in the Prevention of Thromboembolic Events in Patients With Atrial Fibrillation
Brief Title: Evaluating the Use of SR34006 Compared to Warfarin or Acenocoumarol in Patients With Atrial Fibrillation (AMADEUS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EFC5134; SR34006
Record Dates: First submitted 2003-10-06; First posted 2003-10-09 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — idraparinux; Injections; Warfarin; Acenocoumarol; Tablets

INTERVENTIONS:
Drug: SR34006 (idraparinux sodium) Injection
Drug: vitamin K antagonist (warfarin or acenocoumarol) tablets

SUMMARY:
This trial will include patients who have a heart condition called atrial fibrillation. Atrial fibrillation is an abnormal rhythm (irregular beat) in the heart. Patients with atrial fibrillation have an increased chance for a blood clot to form in the heart and move to other blood vessels in the body and cause obstruction. This obstruction may damage tissue. For example, a blood clot plugging a vessel in the brain could cause a stroke. Therefore, patients with atrial fibrillation may be given anticoagulant (blood-thinning) tablets such as warfarin or acenocoumarol.

The purpose of this study is to compare the safety and effectiveness of a new injectable anticoagulant drug that is administered once weekly, SR34006 with warfarin or acenocoumarol tablets.

Assignment to either SR34006 Injection or vitamin K antagonist (warfarin or acenocoumarol) tablets will be purely by chance and will be known by both patients and their doctors.

ELIGIBILITY:
Inclusion Criteria:

* ECG-documented atrial fibrillation (AF) and an indication for long-term vitamin K antagonist (VKA) therapy based on the presence of at least one of the following risk factors:

  1. previous ischemic stroke, transient ischemic attack (TIA) or systemic embolism
  2. hypertension requiring drug treatment
  3. left ventricular dysfunction (left ventricular ejection fraction <45% or symptomatic congestive heart failure)
  4. age >75 years
  5. age between 65-75 years plus diabetes mellitus, or
  6. age between 65-75 years plus symptomatic coronary artery disease (previous myocardial infarction (MI) or angina pectoris)
* Written informed consent

Exclusion Criteria:

* Legal lower age limitations (country specific)
* Indication for VKA other than AF, including prosthetic heart valves, venous thromboembolism, and planned cardioversion
* Transient AF caused by a reversible disorder
* Active bleeding or high risk of bleeding
* Recent (<15 days) or anticipated invasive procedures with potential for uncontrolled bleeding, including major surgery
* Participation in another pharmacotherapeutic study within the prior 30 days
* Creatinine clearance <10 mL/min, severe hepatic disease, or bacterial endocarditis
* Uncontrolled hypertension: systolic blood pressure > 180 mm Hg and/or diastolic blood pressure > 110 mm Hg
* Pregnancy or childbearing potential without proper contraceptive measures
* Breastfeeding
* Any other contraindication listed in the labeling of warfarin or acenocoumarol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4673 (Actual)
Dates: Start 2003-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Composite of all strokes and non-CNS systemic embolism.

SECONDARY OUTCOMES:
Separate components of the primary study outcome.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (84):
- United States (41):
  - Cardiology, P.C., Birmingham, Alabama
  - Oracle Research, a Division of: The Heart Center, P.C., Huntsville, Alabama
  - Arizona Heart Institute Mesa, Mesa, Arizona
  - Saguaro Clinical Research, Tucson, Arizona
  - Southern Arizona Veterans Affairs Health Care System, Tucson, Arizona
  - Office of Dr. Bowden, D.O., Healdsburg, California
  - Jerry L. Pettis VA Medical Center, Loma Linda, California
  - Kenneth W. Carr, M.D. Cardiology, Oceanside, California
  - Richard A. Levy, M.D., San Francisco, California
  - Cardiology Specialists of Orange County, Santa Ana, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Denver Health and Hospital Authority Adult Medicine Clinic, Denver, Colorado
  - Denver Health and Hospital Authority Eastside Health Clinic, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Florida Arrhythmia Consultants, Fort Lauderdale, Florida
  - North Broward Hospital District Cardiovascular Research Institute, Fort Lauderdale, Florida
  - Jacksonville Cardiovascular Clinic, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Wellington Green Family Practice, Wellington, Florida
  - Beacon Medical Research, Indianapolis, Indiana
  - Heart & Vascular Clinic/Advanced Medical Research, Covington, Louisiana
  - The Clinic (Lake Charles Medical & Surgical Clinic), Lake Charles, Louisiana
  - IMG Healthcare, LLC, New Orleans, Louisiana
  - Baystate Medical Center, Springfield, Massachusetts
  - New Mexico Heart Institute, PA, Albuquerque, New Mexico
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Practice of James A. Underberg @ Murray Hill Medical Group, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Oregon Health and Science University, Portland, Oregon
  - Blackstone Cardiology Associates, P.C., Pawtucket, Rhode Island
  - Austin Heart, P.A., Austin, Texas
  - Cardiovascular Research Institute of Dallas, Inc./Cardiology and Internal Medicine Associates, Dallas, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Physicians Office Building (POB), Salt Lake City, Utah
  - McGuire VA Medical Center, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Inland Cardiology, Spokane, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
  - St. Joseph's Hospital, Marshfield, Wisconsin
- Australia (3):
  - Bondi Junction, Cairns, Camperdown, Miranda, Perth
  - Concord Repartiation General Hospital, Concord
  - South Australia, Tasmania, Victoria
- Canada (15):
  - Cardiology Consultant's Group, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Heart Health Institute, Calgary, Alberta
  - University of Calgary, Calgary, Alberta
  - Dr. M.P.J. Senaratne Professional Corporation, Edmonton, Alberta
  - West Coast Cardiology Research, New Westminster, British Columbia
  - Cardiac Arrhythmia Trials, Victoria, British Columbia
  - Health Care Corporation of St. John's Health Sciences Centre, St. John's, Newfoundland and Labrador
  - Zoom International Inc., Saint-Jérôme, Quebec
  - Moose Jaw Cardiac Centre, Moose Jaw, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Saskatoon Medical Specialists, Saskatoon, Saskatchewan
  - Specialists Internal Medicine, Saskatoon, Saskatchewan
  - Dr. Joesph J. Javier, Yorkton, Saskatchewan
  - Yorkton Regional Health Centre, Yorkton, Saskatchewan
- Denmark (3):
  - Faaborg, Fredericia, Frederiksberg, Frederikshavn, Hellerup
  - Herlev, Hillerod, Holstebro, Horsens, Kalundborg, Kobenhavn
  - Kolding, Nykobing Mors, Odense, Skive, Svendborg
- France (3):
  - Bourg En Bresse, Dreux, Lille, Marseille, Maubeuge, Mulhouse
  - Nantes, Nice, Paris, Poitiers, Rennes, Saint Denis
  - Saint-Etienne, Toulouse
- Italy (8):
  - A.O. "Instituti Ospitalieri di Cremona", Cremona
  - Merate, Milano, Padova, Pavia, Piacenza, Reggio Emilia
  - Azienda Ospedaliera San Paolo, Milan
  - Azienda Ospedaliera di Parma, Parma
  - U.O. di Medicina Interna II, Parma
  - Centro Emostasi e Trombosi, Rimini
  - Torino, Treviso
  - Varese
- Netherlands (4):
  - Almelo, Amersfoort, Breda, Boxmeer, Delft, Dordrecht
  - Eindhoven, Enschede, Gorinchem, Gouda, Groningen, Harderwijk
  - Heerlen, Hilversum, Rotterdam, Sneek, Spijkenisse, Tiel
  - Academisch Ziekenhuis Maastricht, Maastricht
- Auckland, Christchurch, Hastings, New Zealand
- Kielce, Krakow, Opole, Plock, Siedlce, Warszawa, Wroclaw, Poland
- United Kingdom (5):
  - University Hospital of Wales, Cardiff
  - Exeter, Dundee, Glasgow, Merseyside, Wirral
  - University of Glasgow, Glasgow
  - Freeman Hospital, Newscastle Upon Tyne
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Ding WY, Lip GYH, Shantsila A. Relationship between Chronic Kidney Disease, Time-in-Therapeutic Range, and Adverse Outcomes in Atrial Fibrillation: A post hoc Analysis from the AMADEUS Trial. Cerebrovasc Dis. 2022;51(1):29-35. doi: 10.1159/000517608. Epub 2021 Jul 28. PMID 34320504
- [Derived] Prins MH, Guillemin I, Gilet H, Gabriel S, Essers B, Raskob G, Kahn SR. Scoring and psychometric validation of the Perception of Anticoagulant Treatment Questionnaire (PACT-Q). Health Qual Life Outcomes. 2009 Apr 7;7:30. doi: 10.1186/1477-7525-7-30. PMID 19348685
- [Derived] Amadeus Investigators; Bousser MG, Bouthier J, Buller HR, Cohen AT, Crijns H, Davidson BL, Halperin J, Hankey G, Levy S, Pengo V, Prandoni P, Prins MH, Tomkowski W, Torp-Pedersen C, Wyse DG. Comparison of idraparinux with vitamin K antagonists for prevention of thromboembolism in patients with atrial fibrillation: a randomised, open-label, non-inferiority trial. Lancet. 2008 Jan 26;371(9609):315-21. doi: 10.1016/S0140-6736(08)60168-3. PMID 18294998
- See also: Related Info — http://www.sanofi-aventis.com